CLINICAL TRIAL: NCT07327931
Title: Comparison of Three Variants of PENG Block Using 20 mL of 0.2% Ropivacaine With Different Combinations of Dexamethasone and Perineural Dexmedetomidine in Patients Aged 65 Years and Older Undergoing Hip Surgery: A Randomized Controlled Trial.
Brief Title: PENG Block Variants With Dexamethasone and Dexmedetomidine in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4/2025
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis; Hip Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG Block With Intravenous Dexamethasone (Active Comparator): Participants will receive a Pericapsular Nerve Group (PENG) block using 20 mL of 0.2% ropivacaine. As part of the study medications, they will receive 4 mg of dexamethasone intravenously and perineural normal saline as placebo, so that the number and volume of injections are identical across all groups.
  Interventions: Drug: Dexamethasone (intravenous)
- PENG Block With Perineural Dexmedetomidine and Intravenous Dexamethasone (Active Comparator): Participants will receive a PENG block using 20 mL of 0.2% ropivacaine combined with 25 µg of dexmedetomidine administered perineurally. In addition, they will receive 4 mg of dexamethasone intravenously. Perineural normal saline may be added to match the total volume of perineural injectate across groups.
  Interventions: Drug: Dexamethasone (intravenous) with Dexmedetomidine (perineural)
- PENG Block With Perineural Dexmedetomidine and Perineural Dexamethasone (Experimental): Participants will receive a PENG block using 20 mL of 0.2% ropivacaine combined with 25 µg of dexmedetomidine and 4 mg of dexamethasone administered perineurally. Intravenously they will receive normal saline as placebo instead of dexamethasone in order to maintain blinding.
  Interventions: Drug: Dexamethasone (perineural) with Dexmedetomidine (perineural)

INTERVENTIONS:
Drug: Dexamethasone (intravenous) — Perineural: 20 mL 0.2% ropivacaine + perineural placebo (normal saline) Intravenous: 4 mg dexamethasone + matching volume of saline if needed
  Arms: PENG Block With Intravenous Dexamethasone
Drug: Dexamethasone (intravenous) with Dexmedetomidine (perineural) — Perineural: 20 mL 0.2% ropivacaine + 25 µg dexmedetomidine (± saline to equalize volume) Intravenous: 4 mg dexamethasone
  Arms: PENG Block With Perineural Dexmedetomidine and Intravenous Dexamethasone
Drug: Dexamethasone (perineural) with Dexmedetomidine (perineural) — Perineural: 20 mL 0.2% ropivacaine + 25 µg dexmedetomidine + 4 mg dexamethasone Intravenous: placebo (0.9% normal saline)
  Arms: PENG Block With Perineural Dexmedetomidine and Perineural Dexamethasone

SUMMARY:
This study will compare three different versions of the Pericapsular Nerve Group (PENG) block in adults aged 65 years and older who are undergoing surgery for hip conditions. The PENG block is a regional anesthesia technique that can reduce pain after surgery and decrease the need for strong opioid pain medications.

All patients in the study will receive the PENG block with 20 mL of 0.2% ropivacaine, but they will be divided into three groups based on the additional medications used:

Group 1: PENG block with ropivacaine plus 4 mg of dexamethasone given intravenously.

Group 2: PENG block with ropivacaine plus 25 micrograms of dexmedetomidine given near the nerves and 4 mg of dexamethasone given intravenously.

Group 3: PENG block with ropivacaine plus 25 micrograms of dexmedetomidine and 4 mg of dexamethasone given near the nerves.

Both dexmedetomidine and dexamethasone are medications that may improve the strength and duration of nerve blocks.

The main goal of this study is to determine which combination provides the best pain control after hip surgery, reduces the need for opioid medications, and improves patient comfort and recovery. We also aim to evaluate the safety and side-effects of each technique.

We hypothesize that adding both dexmedetomidine and dexamethasone near the nerves will provide the longest and most effective pain relief when compared to intravenous administration alone.

This trial may help identify the most effective PENG block formula for older adults undergoing hip surgery and could improve pain management, decrease complications related to opioids, and support faster recovery.

DETAILED DESCRIPTION:
Hip surgery in older adults is commonly associated with significant postoperative pain. Effective pain control is very important in this population because poorly controlled pain may lead to complications such as delayed rehabilitation, increased opioid use, delirium, and longer hospital stay. The Pericapsular Nerve Group (PENG) block is a modern regional anesthesia technique that targets nerves responsible for hip pain while preserving muscle strength around the hip. This may help patients recover faster and walk earlier after surgery.

Dexamethasone and dexmedetomidine are medications that may increase the duration and quality of nerve blocks. Dexamethasone can be given either intravenously or near the nerves. Dexmedetomidine can also be given near the nerves in low doses to prolong pain relief. However, it is still unknown which combination of these medications with the PENG block provides the best results for older patients.

This study will compare three different versions of the PENG block in patients aged 65 years and older who are undergoing hip surgery. All participants will receive 20 mL of 0.2% ropivacaine. They will then be randomly assigned to one of three groups depending on the additional medications they receive:

Group 1: PENG block with 4 mg of dexamethasone given intravenously. Group 2: PENG block with 25 micrograms of dexmedetomidine given near the nerves and 4 mg of dexamethasone given intravenously.

Group 3: PENG block with 25 micrograms of dexmedetomidine and 4 mg of dexamethasone given near the nerves.

The main goal of the study is to determine which combination provides the most effective pain control after surgery. Pain intensity, opioid consumption, side effects, block duration, and time to first mobilization will be measured. The study will also assess safety, possible complications, and patient satisfaction.

We hypothesize that the combination of perineural dexmedetomidine and perineural dexamethasone will result in the longest duration of pain relief with minimal side effects and reduced need for opioids, when compared with intravenous administration.

This is a randomized controlled clinical trial. All patients will receive standard perioperative care. Participation in the study includes follow-up assessments after surgery to evaluate pain levels, medication requirements, and recovery.

The results of this trial may help identify the best regimen for the PENG block in older adults, improve postoperative pain management, reduce opioid-related complications, and support safer and faster rehabilitation after hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Scheduled for elective or emergency hip surgery (e.g., hip fracture fixation or hip arthroplasty)
* ASA physical status I-III
* Ability to communicate pain intensity using the NRS scale
* Written informed consent obtained from the patient or legal representative
* Planned use of PENG block as part of multimodal perioperative analgesia

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* Allergy, intolerance, or contraindication to any study medication: ropivacaine, dexamethasone, dexmedetomidine
* Pre-existing neurological deficit or neuropathy of the affected limb
* Coagulopathy (INR >1.5, platelets <100,000/µL) or current therapeutic anticoagulation that contraindicates regional anesthesia
* Infection at or near the injection site
* Severe hepatic or renal impairment
* History of chronic opioid use (daily opioids >30 days before surgery)
* Cognitive impairment or delirium precluding reliable pain assessment
* BMI > 40 kg/m² (if you want to exclude for technical difficulty)
* Patients receiving another regional nerve block for hip surgery
* Pregnancy or breastfeeding
* Participation in another interventional clinical trial within 30 days

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to First Rescue Analgesia | Within 48 hours after the end of surgery
  Time (in hours) from the end of the PENG block (completion of local anesthetic injection) to the first administration of rescue analgesia (opioid or non-opioid) given for pain intensity ≥4 on the 0-10 Numerical Rating Scale (NRS). Data will be collected from anesthesia records and postoperative medication charts.

SECONDARY OUTCOMES:
Pain Intensity at Rest (NRS 0-10) | 4 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 8 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 12 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 24 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity at Rest (NRS 0-10) | 48 hours after surgery
  Pain intensity at rest assessed using the 0-10 Numerical Rating Scale (0 = no pain, 10 = worst imaginable pain). Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 4 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 8 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 12 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 24 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Pain Intensity During Movement (NRS 0-10) | 48 hours after surgery
  Pain intensity during standardised hip movement (e.g., flexion or assisted mobilization) assessed using the 0-10 Numerical Rating Scale. Mean NRS scores at each time point will be compared between groups.
Total Opioid Consumption | 0-48 hours after surgery
  Cumulative dose of all opioid analgesics administered in the postoperative period, converted to oral morphine milligram equivalents (MME). Values at 24 and 48 hours will be recorded and compared between groups.
Incidence of Postoperative Nausea and Vomiting (PONV) | 0-48 hours after surgery
  Presence of nausea and/or vomiting requiring antiemetic therapy. The proportion of patients with at least one episode of PONV will be recorded and compared between groups
Hemodynamic Adverse Events (Hypotension and Bradycardia) | From block placement until 24 hours after surgery
  Incidence of hypotension (e.g., systolic blood pressure <90 mmHg or decrease >30% from baseline) and bradycardia (heart rate <50 beats/min) requiring medical treatment. Events will be recorded and compared between groups.
Block-Related Adverse Events, Including Neurological Complications | From block placement until hospital discharge, up to 30 days
  Incidence of complications potentially related to the PENG block or perineural adjuvants, including signs of local anesthetic systemic toxicity, prolonged motor or sensory deficit, nerve injury (evaluated in the postoperative clinic or outpatient nerve injury clinic if required), infection at the injection site, hematoma, or persistent weakness.
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 4 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 8 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 12 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 24 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia
Motor Function Preservation (Quadriceps Strength, MRC Scale) | 48 hours after surgery
  Quadriceps muscle strength will be evaluated using the Medical Research Council (MRC) scale, ranging from 0 (no contraction) to 5 (normal power), at 4, 8, 12, 24, and 48 hours to detect any motor impairment associated with the applied regional anesthesia 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications arising from this study will be made available to qualified researchers upon reasonable request. Shared data will include baseline characteristics, outcome measures, and safety data necessary to reproduce the main analyses. All data will be fully anonymized prior to sharing to protect participant privacy.
Time Frame: The data will become available beginning 6 months after publication of the primary results and will remain available for 5 years following publication.
Access Criteria: Access to the data will be granted to researchers who provide a methodologically sound research proposal. Requests must be approved by the principal investigator and the local ethics committee, if required. Data will be shared under a data use agreement and may be used only for non-commercial scientific research purposes.